CLINICAL TRIAL: NCT00283218
Title: A Comparison of Pharmacodynamics and Pharmacokinetics of Insulin Aspart, Biphasic Insulin Aspart 30, 50 and 70. - A Randomised, Quadruple Cross-Over Trial
Brief Title: A Comparison of Pharmacodynamics and Pharmacokinetics of Insulin Aspart, Biphasic Insulin Aspart 30, 50 and 70.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Asp-BIAsp-2005/0109
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2006-08-08 (Estimated); Status verified 2006-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

INTERVENTIONS:
Drug: NovoRapid, NovoMix 30, Bifasisk Insulin Aspart 50, BIAsp70

SUMMARY:
The hypothesis is that an optimal formulation of fast acting and intermediary acting insulin analogues will improve post prandial glycaemic control in patients with type 1 diabetes.

OBJECTIVE:

The objective is to describe pharmacodynamic (PD) and pharmacokinetic (PK) profiles of Insulin Aspart (IAsp), Biphasic Insulin Aspart (BIAsp) 30, 50 and 70 for a period of 12 hours following a standard test meal on four days respectively in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
This trial is a single centre, open-label, randomised 4 period cross-over trial, comparing the pk and pd profiles of IAsp, BIAsp 30, BIAsp 50 and BIAsp 70 after a standard test meal in subjects with type 1 diabetes. The profiles will be derived over a 12-hour period after subcutaneous injection in the abdominal region with a single dose of IAsp, BIAsp 30, BIAsp 50 or BIAsp 70 at a test meal. The trial consists of a screening period of 4-21 days and 4 treatment visits

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities.
2. Diagnosed type 1 diabetes before the age of 40 and on insulin treatment within one year of diagnosis.
3. Insulin treatment of any regime for more than one year at time of inclusion.
4. Total insulin demand ≥ 0,5 IU/kg/24 hrs
5. HbA1c between 7% and 12 % (both values included).
6. Age ≥ 18 years.
7. BMI between 18 and 35 kg /m2 (including both values).

Exclusion Criteria:

1. Known or suspected allergy to trial product(s) or related products.
2. Recurrent major hypoglycaemic episodes.
3. Heart: Unstable Angina Pectoris, AMI < 12 months or heart insufficiency classified according to NYHA III-IV
4. Blood Pressure: Severe uncontrolled hypertension with BP > 180/110 mmHg, sitting
5. Liver: Impaired hepatic function corresponding to serum-ALAT or -basic phosphatase > 2x upper reference limit of the local laboratory.
6. Kidneys: Impaired renal function corresponding to serum-creatinin > 150 μmol/l according to the local laboratory.
7. Any disease judged by the investigator to affect the trial.
8. Pregnancy, breast feeding or the intention of becoming pregnant or fertile women not using adequate contraceptive measures - adequate contraceptive method is sterilisation, hysterectomy or current use of contraceptive pills or intra uterine device.
9. The receipt of any investigational drug within a three month period prior to this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Primary endpoint:
• Cmaxglu: Peak plasma glucose following test meal (breakfast). A comparison will be made between BIAsp 50 vs BIAsp 70, BIAsp 30 vs BIAsp 70, BIAsp 30 vs BIAsp 50 and IAsp vs BIAsp 30, 50 and 70.

SECONDARY OUTCOMES:
Secondary endpoints:
AUCglu: The area under the plasma glucose concentration (0-12, 0-6, 6-12, 0-4, 4-8, 8-12 hours after test meal) after a single injection of one of the four insulin aspart preparation: IAsp (NovoRapid®), Biphasic insulin aspart 30, 50 and 70.
AUCins: The area under insulin aspart concentration (0-12, 0-6, 6-12, 0-4, 4-8, 8-12 hours after test meal) after a single injection of one of the four insulin aspart preparation: IAsp (NovoRapid®), Biphasic insulin aspart 30, 50 and 70.

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christiansen, M.D., Principal Investigator — Medicinsk Afd. M, Århus Sygehus, Nørrebrogade 44, 8000 Århus C; Tina Parkner, M.D., Study Director — Medicinsk Afd. M, Århus Sygehus, Nørrebrogade 44, 8000 Århus C; Niels Ejskjaer, M.D., Study Director — Medicinsk afd. M, Århus Sygehus, Nørrebrogade 44, 8000 Århus C; Rannveig L Thorisdottir, Stud.med, Study Director — Medicinsk afd. M, Århus Sygehus, Nørrebrogade 44, 8000 Århus C
Locations (1):
- Dept of Medicine M, Aarhus University Hospital, Nørrebrogade 44, Aarhus, C, Denmark

REFERENCES:
- [Background] Weyer C, Heise T, Heinemann L. Insulin aspart in a 30/70 premixed formulation. Pharmacodynamic properties of a rapid-acting insulin analog in stable mixture. Diabetes Care. 1997 Oct;20(10):1612-4. doi: 10.2337/diacare.20.10.1612. PMID 9314644
- [Background] Jacobsen LV, Sogaard B, Riis A. Pharmacokinetics and pharmacodynamics of a premixed formulation of soluble and protamine-retarded insulin aspart. Eur J Clin Pharmacol. 2000 Aug;56(5):399-403. doi: 10.1007/s002280000159. PMID 11009049
- [Background] Kang S, Creagh FM, Peters JR, Brange J, Volund A, Owens DR. Comparison of subcutaneous soluble human insulin and insulin analogues (AspB9, GluB27; AspB10; AspB28) on meal-related plasma glucose excursions in type I diabetic subjects. Diabetes Care. 1991 Jul;14(7):571-7. doi: 10.2337/diacare.14.7.571. PMID 1914797
- [Background] Boehm BO, Home PD, Behrend C, Kamp NM, Lindholm A. Premixed insulin aspart 30 vs. premixed human insulin 30/70 twice daily: a randomized trial in Type 1 and Type 2 diabetic patients. Diabet Med. 2002 May;19(5):393-9. doi: 10.1046/j.1464-5491.2002.00733.x. PMID 12027927